CLINICAL TRIAL: NCT06333548
Title: Comparison of Cord Blood Alarin Levels in Term Babies According to Birth Weight
Brief Title: Cord Blood Alarin Levels in Term Babies
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Melek Buyukeren, Associate Professor, Konya City Hospital
Other Study IDs: KSH_MB_2024_1
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Birth Weight
Keywords: NEWBORN; ALARİN; UMBİLİCAL CORD BLOOD
MeSH Terms: conditions — Birth Weight | interventions — Gestational Age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Appropriate for gestational age: Appropriate for gestational age
  Interventions: Diagnostic Test: Appropriate for gestational age , small for gestational age, large for gestational age, Baby of mother diagnosed with GDM
- small for gestational age: small for gestational age
  Interventions: Diagnostic Test: Appropriate for gestational age , small for gestational age, large for gestational age, Baby of mother diagnosed with GDM
- large for gestational age: large for gestational age
  Interventions: Diagnostic Test: Appropriate for gestational age , small for gestational age, large for gestational age, Baby of mother diagnosed with GDM
- Baby of mother diagnosed with GDM: Baby of mother diagnosed with gestational diabetes mellitus
  Interventions: Diagnostic Test: Appropriate for gestational age , small for gestational age, large for gestational age, Baby of mother diagnosed with GDM

INTERVENTIONS:
Diagnostic Test: Appropriate for gestational age , small for gestational age, large for gestational age, Baby of mother diagnosed with GDM — No intervention

SUMMARY:
In this study, alarin levels in the cord blood of babies with large birth weights will be compared with babies of normal weight. Thus, the investigators aimed to find out whether there is a relationship between babies' birth weights and alarin.

DETAILED DESCRIPTION:
Studies have shown that the galanin neuropeptide family plays a role in regulating appetite, insulin resistance, obesity, hypertension and metabolism. Alarin is a peptide consisting of 25 amino acids. Current research shows that allerin plays an important role in the emergence and development of diabetes and obesity. There are studies that found that the serum alarin level increased significantly in patients with impaired glucose tolerance and type 2 diabetes mellitus. Additionally, studies have found that both non-obese and obese type 2 diabetes mellitus serum alarin levels increase.

Studies in the literature are related to adults, and there are no studies on alarin levels in newborn babies.

Based on the alarin studies available in the literature, the investigators determined whether there is a relationship between the alarin level and the baby's birth weight by comparing the alarin level in the cord blood of babies with a high birth weight according to their gestational age (both babies of diabetic mothers and babies of non-diabetic mothers) compared to babies whose birth weight is within the normal range. the investigators aimed to find it.

ELIGIBILITY:
Inclusion Criteria:

* Babies given consent by their families
* Healthy babies

Exclusion Criteria:

* Babies with syndromic appearance or any accompanying disease
* Babies whose family does not give consent

Ages: 1 Minute to 5 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies born between the planned dates and whose families gave consent for the study were divided into four different groups according to their characteristics:
  1. Babies with normal weight according to gestational age (AGA): 25 babies were included in the study.
  2. Low weight babies for gestational age (SGA): 20 babies were included in the study.
  3. Large-weight babies for gestational age (LGA): 22 babies were included in the study.
  4. Babies whose mothers had gestational diabetes mellitus: 20 babies were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Comparison of cord blood alarin levels of babies in different groups according to birth weight (low-appropriate-large) and babies of mothers diagnosed with gestational diabetes regardless of birth weight. | postnatal 5 minutes
  umbilical cord blood alarin levels

CONTACTS AND LOCATIONS:
Overall Officials: MELEK BUYUKEREN, Study Director — Konya City Hospital
Locations (1):
- MELEK, Konya, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan and Clinical Study Report
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months after the article was published
Access Criteria: The data set generated and analyzed in this study are available from corresponding author on a reasonable request.

REFERENCES:
- [Result] Zhou X, Luo M, Zhou S, Cheng Z, Chen Z, Yu X. Plasma Alarin Level and Its Influencing Factors in Obese Newly Diagnosed Type 2 Diabetes Patients. Diabetes Metab Syndr Obes. 2021 Jan 27;14:379-385. doi: 10.2147/DMSO.S290072. eCollection 2021. PMID 33536771
- [Result] Hu W, Fan X, Zhou B, Li L, Tian B, Fang X, Xu X, Liu H, Yang G, Liu Y. Circulating alarin concentrations are high in patients with type 2 diabetes and increased by glucagon-like peptide-1 receptor agonist treatment: An Consort-compliant study. Medicine (Baltimore). 2019 Jul;98(28):e16428. doi: 10.1097/MD.0000000000016428. PMID 31305464